CLINICAL TRIAL: NCT01254968
Title: Influence of Direction of Movement While Walking Upon the Blood Flow Rate Through Brain, Examined by Transcranial Doppler Sonography in Young Healthy Subjects.
Brief Title: Influence of Direction of Movement While Walking
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Medical University of Silesia, Department of Rehabilitation
Other Study IDs: BW-07-AM
Record Dates: First submitted 2010-11-29; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-11

CONDITIONS: Changes in Blood Flow to the Brain; Changes Depending on the Form of Walking
Keywords: blood flow in the middle cerebral artery of brain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- examining group: 20 healthy subjects (11 men, 9 women, average age 23.94)
- control group: 6 healthy subjects (3 men, 3 women, average age 23.6)

SUMMARY:
The aim of the study is evaluation of cerebral blood flow (based on testing the rate of flow in middle cerebral arteries by transcranial Doppler ultrasound) during different forms of walking training - walk forwards and backwards, with closed and open eyes.

DETAILED DESCRIPTION:
In the third minute of training walking a significant increase in blood flow velocity was recorded, both in right and left middle cerebral arteries. It was observed in the left artery during all forms of training. In the right artery it occurred only during three forms of difficult training, and was preceded by significant decrease in blood flow in the first minute of the gait with eyes closed. The output values of the rate of blood flow in both right and left middle cerebral arteries became progressively reduced in the successive stages of gait. Pressure and pulse rates did not correlate with the variables of blood flow velocity in middle cerebral arteries.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects without brain disease

Exclusion Criteria:

* brain disease and walking disfunctions

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 healthy subjects (11 men, 9 women, average age 23.94) participated in a study measuring the speed of blood flow in middle cerebral arteries using transcranial Doppler (transcranial Doppler Sonography) while walking on a treadmill.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-12; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Transcranial Doppler sonography in young healthy subjects. | 5 months
  Significant changes in blood flow to the brain depending on the form of walking and its conditions were observed. Changes in the right middle cerebral artery were more diverse than in the left artery. Difficulty in walking training forms gave long-term vasodilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Silesia, Katowice, Silesian Voivodeship, Poland